CLINICAL TRIAL: NCT04698018
Title: A Trial Investigating the Pharmacokinetic Properties of Fast-acting Insulin Aspart in Chinese Subjects With Type 1 Diabetes or Type 2 Diabetes
Brief Title: A Research Study to Look at How Faster Aspart Works in Chinese People With Type 1 Diabetes or Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1218-4316; U1111-1199-1934 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-12-21; First posted 2021-01-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Faster aspart (Experimental): Subjects will receive 2 injections of a single dose of faster aspart at a predefined fixed dose level (0.2 U/kg body weight) for type 1 diabetes and (0.3 U/kg body weight) if subject has type 2 diabetes.
  Interventions: Drug: Faster Aspart
- NovoRapid® (Active Comparator): Subjects will receive 2 injections of a single dose of NovoRapid® at a predefined fixed dose level (0.2 U/kg body weight) for type 1 diabetes and (0.3 U/kg body weight) if subject has type 2 diabetes.
  Interventions: Drug: Novo Rapid

INTERVENTIONS:
Drug: Faster Aspart — Administered s.c. (subcutaneously, under the skin) of the lower abdomen using a pen-injector.
  Arms: Faster aspart
Drug: Novo Rapid — Administered s.c. (subcutaneously, under the skin) of the lower abdomen using a pen-injector.
  Arms: NovoRapid®

SUMMARY:
This study looks at how faster aspart reaches and stays in the blood after injection in Chinese people with type 1 diabetes or type 2 diabetes, compared to the reference product called NovoRapid®. Participants will get both faster aspart and NovoRapid®. The order in which Participants get them is decided by chance. Participants will get each study medicine once during the study meaning that they will get a total of 2 injections with study medicines. The medicine will be injected under the skin of the lower abdomen. The study will last for about 19-72 days. Participants will have 5 clinic visits with the study doctor (including the one in which participants give their consent). Participants will need to stay overnight for 2 of the 5 clinic visits. Participants will have blood samples taken during some of the clinic visits. During the visits where participants get the study medicines, samples of their blood will be taken several times for up to 12 hours after getting the study medicine.

ELIGIBILITY:
Inclusion criteria:

For a subject with type 1 diabetes mellitus:

* Male or female Chinese subjects aged 18-64 years (both inclusive) at the time of signing informed consent.
* Type 1 diabetes mellitus (as diagnosed clinically) greater than or equal to 12 months prior to the day of screening.
* Treated with multiple daily insulin injections or premix insulin greater than or equal to 12 months prior to the day of screening or treated with continuous subcutaneous insulin infusion (CSII) greater than or equal to 3 months prior to the day of screening.
* Glycosylated haemoglobin (HbA1c) less than or equal to 9.0 percent (75 mmol/mol) by central laboratory analysis.

For a subject with type 2 diabetes mellitus:

* Male or female Chinese subjects aged 18-75 years (both inclusive) at the time of signing informed consent.
* Type 2 diabetes mellitus (as diagnosed clinically) greater than or equal to 12 months prior to the day of screening.
* Treated with multiple daily insulin injections or premix insulin greater than or equal to 6 months prior to the day of screening or treated with continuous subcutaneous insulin infusion (CSII) greater than or equal to 3 months prior to the day of screening.
* Glycosylated haemoglobin less than or equal to 9.5 percent (80 mmol/mol) by central laboratory analysis.

Exclusion criteria:

For a subject with type 1 diabetes mellitus or type 2 diabetes mellitus:

* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Surgery or trauma with significant blood loss (more than 400 mL) within the last 3 months prior to screening.
* Not able or willing to refrain from smoking and use of nicotine substitute products during the in-patient period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
AUCIAsp,0-30min, area under the serum insulin aspart concentration-time curve from 0 to 30 minutes | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L

SECONDARY OUTCOMES:
AUCIAsp,0-15min, area under the serum insulin aspart concentration-time curve from 0 to 15 minutes | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L
AUCIAsp,0-1h, area under the serum insulin aspart concentration-time curve from 0 to 1 hour | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L
AUCIAsp,0-1½h, area under the serum insulin aspart concentration-time curve from 0 to 1½ hours | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L
AUCIAsp,0-2h, area under the serum insulin aspart concentration-time curve from 0 to 2 hours | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L
AUCIAsp,0-12h, area under the serum insulin aspart concentration-time curve from 0 to 12 hours | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol·h/L
Cmax,IAsp, maximum observed serum insulin aspart concentration | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  pmol/L
tmax,IAsp, time to maximum observed serum insulin aspart concentration | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  Minutes
Onset of appearanceIAsp, time from trial product administration until the first time serum insulin aspart concentration greater than or equal to lower limit of quantification (LLOQ) | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  Minutes
Time to 50 percent Cmax, IAsp, the first time point where the insulin aspart concentration equals 50 percent of Cmax,IAsp | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  Minutes
Time to late 50 percent Cmax,IAsp, the last time point where the insulin aspart concentration equals 50 percent of Cmax,IAsp | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  Minutes
t½, terminal half-life for insulin aspart | 0 to 12 hours after dosing on Day 2 of Visit 2 (3-21 days after screening) and Visit 3 (7-28 days after visit 2, day 2)
  Minutes
Number of treatment emergent adverse events | Until 7 days after IMP (investigational medicinal product) administration
  Count of Events
Number of treatment emergent hypoglycaemic episodes | No longer than 16 hours after IMP administration until next administration of insulin (non-investigational medicinal product (NIMP) or subject's pre-trial insulin)
  Count of Episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (3):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
- Hong Kong (2):
  - Phase 1 Clinical Trial Centre, Shatin, New Territories, Hong Kong
  - Phase 1 Clinical Trial Centre, Shatin, New Territories

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com